CLINICAL TRIAL: NCT01581112
Title: Microbial Community Transplantation on the Armpit/Foot in Order to Reduce the Malodour Generation on Armpit/Foot
Brief Title: Microbial Community Transplantation on the Armpit/Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/256
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Heavy, Bad Body Odour From Armpit; Heavy, Bad Body Odour From Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heavy armpit odour (Experimental): Subjects with heavy armpit odour.
  Interventions: Biological: Microbial transplant
- Heavy foot odour (Experimental): Subjects with heavy foot odour.
  Interventions: Biological: Microbial transplant

INTERVENTIONS:
Biological: Microbial transplant — Every subjects has 2 armpits and 2 feet. One armpit/foot is treated, the other is not treated.

SUMMARY:
The malodour generation of a person's armpit/foot is caused by the bacteria thriving on that armpit/foot. In order to alter or reduce once bad body odour or foot odour, the living microbial community on the foot/armpit of a non-malodorous person will be transmitted (or up scaled and transmitted) to the foot/armpit of a malodorous person. The odour is evaluated by a trained smelling panel, the bacteria living on the armpit/foot is examined by means of molecular techniques. The microbial transplantation and its follow-up happens under the supervision of a doctor.

ELIGIBILITY:
Inclusion Criteria:

* Bad armpit or foot odour

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in odour severity after bacterial transplantation | Baseline and day 1
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and day 2
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and day 3
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and day 4
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and day 5
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and week 2
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and week 3
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and week 4
  Odour evaluation by a trained smelling panel.
Change in molecular characterisation of the bacterial community. | Baseline and day 1
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and day 2
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and day 3
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and day 4
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and day 5
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and week 2
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and week 3
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community. | Baseline and week 4
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).

SECONDARY OUTCOMES:
Change in odour severity after bacterial transplantation | Baseline and 2 months
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and 4 months
  Odour evaluation by a trained smelling panel.
Change in odour severity after bacterial transplantation | Baseline and 6 months
  Odour evaluation by a trained smelling panel.
Change in molecular characterisation of the bacterial community | Baseline and 2 months
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community | Baseline and 4 months
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).
Change in molecular characterisation of the bacterial community | Baseline and 6 months
  Microbial evaluation by means of DNA extraction and Denaturing Gradient Gel Electrophoresis (DGGE).

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University, Ghent, Belgium